CLINICAL TRIAL: NCT01761669
Title: Does Deficiency in Vitamin D Induced Hypercoagulation or Thrombin Generation
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Elias mazen, Director of Internal Medicine C, HaEmek Medical Center, Israel
Other Study IDs: vitamin D
Record Dates: First submitted 2012-12-04; First posted 2013-01-07 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2014-12

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Vitamin D

STUDY DESIGN:
Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- healthy voulnters
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Vitamin D

SUMMARY:
Working hypothesis and aims: The aim of our study is to investigate whether vitamin D deficiency could cause increased thrombin generation and a hypercoagulable state healthy volunteers.

Methods:

In total 400 healthy volunteers are planned for inclusion in this trial. After signing an informed consent two blood samples will be obtained from each participant.

Expected results: invastigator expect to find that volunteers with vitamin D deficiency will have thrombin generation curve compatible with hypercoagulable state and returning to normal after treatment with vitamin D

ELIGIBILITY:
Inclusion Criteria: age >18 healthy naive to drug treatment -

Exclusion Criteria:

no exc criteria

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 400 healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2013-04; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
the correlation between vitamin D levels and endogenous thrombin potential | 3 month
  one blood test

CONTACTS AND LOCATIONS:
Overall Officials: mazen elias, MD, Principal Investigator — Emek Medical Center
Locations (1):
- HaEmekMC, Afula, Israel